CLINICAL TRIAL: NCT07135115
Title: Targeting Lifestyle to Improve Colorectal Cancer Screening
Acronym: KoloPrev
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian Institute of Public Health (Other Government)
Collaborators: University of Oslo (Other); Norwegian Cancer Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 572721; 223165 (Other Grant/Funding Number: The Norwegian Cancer Society)
Record Dates: First submitted 2025-08-11; First posted 2025-08-21 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Lifestyle Alteration; Tobacco; Diet Modification; Physical Activity; Alcohol Consumption; Body Weight Control
Keywords: Lifestyle intervention; Colorectal cancer screening; Diet; Alcohol consumption; Smoking; Body mass index; Physical activity; Digital questionnaire
MeSH Terms: conditions — Motor Activity; Alcohol Drinking; Smoking

STUDY DESIGN:
Intervention Model Description: This is a five-armed, parallel group and randomized controlled trial. Three of the arms are intervention arms, while two arms are control arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Lifestyle advice, low intensity (Experimental): The participants will receive digital personally tailored diet and lifestyle advice (the Digikost report) after completion of the Digikost questionnaire at baseline.
  Interventions: Behavioral: Digikost report baseline only
- Lifestyle advice, medium intensity (Experimental): The participants will receive digital personally tailored diet and lifestyle advice (the Digikost report) after completion of the Digikost questionnaire at baseline and after each 6 months through the 2-year intervention period.
  Interventions: Behavioral: Digikost report intensive
- Lifestyle advice, high intensity (Experimental): The participants will receive digital personally tailored diet and lifestyle advice (the Digikost report) after completion of the Digikost questionnaire at baseline and after each 6 months through the 2-year intervention period. Additionally, the participants will be offered an individual telephone counselling meeting on his/her Digikost report with an advisor at baseline, as well as invited to inspirational webinars on cancer preventive lifestyle every 6 months.
  Interventions: Behavioral: Digikost report intensive with individual counselling and webinars
- Control (No Intervention): The participants will be invited to complete the Digikost questionnaire at baseline and after 6 months and 2 years, but will not receive the Digikost report after completing the questionnaire.
- Usual care (No Intervention): Participants will be treated only with the current standard of practice in ColorectalScreen Norway. Participants will not be informed of the trial, invited to fill in the Digikost questionnaire or receive the Digikost report.

INTERVENTIONS:
Behavioral: Digikost report baseline only — The Digikost report will be made available for the participant immediately after completing of the Digikost questionnaire at baseline.
  Arms: Lifestyle advice, low intensity
Behavioral: Digikost report intensive with individual counselling and webinars — The Digikost report will be made available for the participant each time after completion of the Digikost questionnaire every 6 months. Additionally, the participant is offered an individual lifestyle counselling meeting by telephone at baseline and invited to inspirational webinars on cancer preventive lifestyle every 6 months.
  Arms: Lifestyle advice, high intensity
Behavioral: Digikost report intensive — The Digikost report will be made available for the participant each time after completion of the Digikost questionnaire every 6 months.
  Arms: Lifestyle advice, medium intensity

SUMMARY:
The goal of this study is to learn whether receiving personalized, digital lifestyle advice during colorectal cancer screening leeds to changes in lifestyle over a two-year follow-up period. Changes will be measured using a composite score including diet, alcohol consumption, physical activity, body mass index and smoking habits. The main questions it aims to answer are:

* Do participants who receive short, personalized digital feedback on their lifestyle - either once or through repeated rounds -change their lifestyle during the two-year study period, compared to those who do not receive any feedback?
* Does the inclusion of additional contact, such as telephone consultation with healthcare providers, result in further lifestyle changes?

Researchers will compare three groups which receive digital feedback at different intensities and a control group which does not get any feedback to see if lifestyle changes differ between the groups.

Participants in four different groups will fill in a digital diet and lifestyle questionnaire at the start of the study and 2-4 times after this during the following 2 years.

* Participants in three of the groups will receive a short digital feedback report on their lifestyle related to health recommendations after each completion of the questionnaire.
* One of these groups will also be offered to go through the feedback report together with a healthcare provider in a telephone call.
* This group will also receive invitations to motivational webinars every half year during the 2-year study period. The topics in the webinars address cancer preventive lifestyle.

A secondary goal of the study is to understand whether the invitation to fill in the diet and lifestyle questionnaire affects participation in colorectal cancer screening. Therefore, a fifth group of individuals invited to colorectal cancer screening but not to be invited to fill in the questionnaire will be included for extra comparison. Participation in colorectal cancer screening will be compared between this group and the four groups that are additionally invited to complete the questionnaire.

Another secondary goal is to learn which groups in the society consent to the current study. Therefore, sociodemographic characteristics will be compared between the invited individuals who consent and those who do not consent to the study.

DETAILED DESCRIPTION:
This is a five-armed, parallel group randomized controlled trial (RCT) among participants invited to the national colorectal cancer screening programme in Norway (ColorectalScreen Norway). The aim of the trial is to test the effect of intervention with a digital, personally tailored diet and lifestyle feedback (Digikost report) on dietary and lifestyle changes in colorectal cancer screening participants. Additionally, it is an aim to gain knowledge on feasibility and acceptability of the digital diet and lifestyle assessment and feedback at colorectal cancer screening setting.

PRIMARY AIM The main aim is to study the effect of the intervention on 2-year changes in a healthy lifestyle score.

SECONDARY AIMS:

To study:

* the effect of the intervention on 6-month changes in a healthy lifestyle score
* whether the effect on changes in the score is dependent on the intensity of the feedback
* whether introduction of the digital diet and lifestyle questionnaire at ColorectalScreen Norway affects screening participation rate
* participation rate in the digital diet and lifestyle questionnaire, and sociodemographic participant vs. non-participant characteristics
* the perceptions and accept of the digital tool in CRC screening participants.
* feasibility of conducting the study
* cancer incidence, overall mortality and cancer-specific mortality in this study population until year 2040.

RANDOMIZATION AND THE STUDY ARMS The study will randomize a total of 16,000 individuals invited to ColorectalScreen Norway in a defined time period into the following five arms (1:1:1:1:1): three intervention arms (arm A, B and C), a control arm and an arm not receiving an invitation to the study ("usual care", i.e. usual screening service).

A total of 12,800 colorectal cancer screening invitees will be invited to one of the four trial arms (a control arm and three intervention arms, 3,200 invitees in each arm).

The study arms consist of 19 Hospital Trust strata: Finnmark, Helgeland, Innlandet, Førde, Sørlandet, Telemark, Fonna, Ahus, Bergen, Møre og Romsdal, OUS, Vestre Viken, Østfold, Stavanger, Nordland, Vestfold, UNN, St. Olavs and Nord-Trøndelag. As the randomization in this study is stratified, ColorectalScreen Norway invitees are first divided into strata, and then randomly assigned to one of the five arms. The study has a parallel group design, meaning there are no crossovers between the five arms.

INTERVENTION The intervention in this study is digital individually tailored advice to follow the Norwegian food-based dietary guidelines, including recommendations on physical activity, body weight and avoidance of tobacco.

In the three intervention arms (A, B and C), the participants are asked to complete digital assessment of diet and lifestyle (Digikost questionnaire) at different intensities during the 2-year intervention period.

The digital personalized advice (Digikost report) will be made available and sent automatically to the participant's e-mail immediately after completing the Digikost questionnaire. The intervention will last for up to 2 years, with the number of questionnaire rounds and intensity depending on the study arm. The intensities in the three arms will be:

Intervention arm A: Invitation to complete Digikost questionnaire sent at baseline and after 6 months. The digital advice in the Digikost report will be made available for the participant in an e-mail sent immediately after completion of the Digikost questionnaire at baseline, but not after 6 months.

Intervention arm B: Invitation to complete Digikost questionnaire sent at baseline and after each 6 months through the intervention period, in total four times. The digital advice in the Digikost report will be made available for the participant in an e-mail sent immediately after completion of the Digikost questionnaire.

Intervention arm C: Invitation to complete Digikost questionnaire sent at baseline and after each 6 months through the intervention period, in total four times. The digital advice in the Digikost report will be made available for the participant in an E-mail sent immediately after completion of the Digikost questionnaire. At baseline, the participant will additionally be offered an individual consultation telephone meeting with a healthcare provider, scheduled to take place shortly after the baseline assessment. Information of this offer will be given after completion of the questionnaire. Additionally, the participants will be invited, through e-mail, to inspirational webinars on cancer preventive lifestyle every 6 months, with possibilities for submitting questions prior to the seminar.

The Digikost report will be made available for the participants in the intervention arms A, B and C also after the 2-year Digikost questionnaire at the end of the study period. This, however, is not part of the intervention, but rather a reward for the participants.

COMPARATOR The first comparator (the Control arm) will be invited to complete the digital lifestyle questionnaire at baseline, after 6 months and 2 years, but will not receive any feedback. The second comparator (the "Usual care" arm) is the current standard of practice in ColorectalScreen Norway. The Usual care arm will not receive any questionnaire or feedback.

For one of the secondary aims (sociodemographic participant vs. non-participant characteristics), the group of individuals who complete the questionnaire at baseline will be compared with the group of individuals who do not complete the questionnaire.

ENDPOINTS The primary endpoint, for comparison between Intervention arms A, B and C and Control arm is change in a healthy lifestyle score, which consists of the 2018 WCRF/AICR Score and smoking status. This is defined as difference in the score for each participant assessed at baseline and after the 2-year intervention period. The 2018 WCRF/AICR Score is a point score based on the participant's answers in the Digikost questionnaire. Zero to one point is given for the grade to which the participant complies to each of the seven health recommendations: 1) normal body weight, 2) physical activity, 3) diet rich in wholegrains, vegetables, fruit and beans, 4) limited intake of 'fast foods' and other processed foods high in fat, starches or sugars, 5) limited consumption of red and processed meat, 6) limited consumption of sugar-sweetened drinks, and 7) low alcohol consumption. The 2018 WCRF/AICR Score thus ranges from 0 to 7 points. Added by one score point for smoking status, the healthy lifestyle score will range from 0 to 8 points.

SECONDARY ENDPOINTS

* change in the healthy lifestyle score after six months (comparison between the Intervention arms A, B and C and Control arm)
* participation in CRC screening, defined as return of the faecal screening sample at baseline (comparison between the Intervention arms and Control arm, and the Usual care arm)
* participation in the digital lifestyle questionnaire, that is completing the questionnaire at baseline vs. not completing the questionnaire (comparison between different sociodemographic groups)
* attendance in the personal consultation telephone meetings and the motivational webinars, and retention rate
* long-term cancer incidence, total mortality and cancer-specific mortality (comparison between the Intervention arms A, B and C, Control arm and Usual care arm)
* the acceptability and usefulness of the Digikost tool as perceived by the participants (a qualitative sub-study, described further below).

DATA FROM OTHER SOURCES

* Statistics Norway data on sociodemographic characteristics (education level, household number, household income, marital status, cohabitation status, immigration status and country of birth). This is to analyse the characteristics of participants vs. non-participants of the Digikost questionnaire.
* Colorectal cancer screening result at the current and upcoming screening rounds up to five years from invitation to the KoloPrev study, including results from the faecal screening test and colonoscopy findings, drawn from the administrative data system of ColorectalScreen Norway. This is to analyse the intervention effect in more detail, separating between screening participants with 1) positive vs. negative screening test, and 2) precancer and cancer findings, and without screening findings.
* Cancer Registry data on all cancer incidences until Dec 31, 2040. This is to analyse the intervention effect on the long-term hard endpoints, both by intention-to-treat and per-protocol approach.
* Cause of Death Registry data until Dec 31, 2040. This is to analyse the intervention effect on the long-term hard endpoints, both by intention-to-treat and per-protocol approach.

THE QUALITATIVE STUDY In order to determine the acceptability of introducing a rapid lifestyle assessment with personalized feedback into the national CRC screening program, the researchers will perform a formative evaluation.

A longitudinal qualitative study will be conducted among a subsample of the intervention group. Individual interviews using semi-structured interview guides will be used to collect the participant's perceptions of the acceptability of completing the Digikost and receiving personalized feedback within the context of the CRC screening, as well as whether they found the feedback motivating. The participants will be followed-up a month after the first interview to collect their motivation and experiences with implementing any lifestyle changes based on the personalized advice.

ELIGIBILITY:
Inclusion Criteria:

* Invited to the first round of immunochemical faecal blood testing in the national colorectal cancer screening program via a digital platform.

Exclusion Criteria:

* Not invited to the national colorectal cancer screening program.

Ages: 55 Years to 56 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16000 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2028-05-31 (Estimated); Study Completion 2041-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in a healthy lifestyle score | From baseline to the end of intervention at 24 months
  Difference in a healthy lifestyle score, which consists of the 2018 WCRF/AICR Score added by smoking status for each participant, assessed at baseline and after the 2-year trial period. The healthy lifestyle score is a point score based on the participant's answers in the lifestyle questionnaire. 0-1 point is given for the grade to which the participant complies to each of the eight health recommendations: 1) normal body weight, 2) physical activity, 3) diet rich in wholegrains, vegetables, fruit and beans, 4) limited intake of 'fast foods' and other processed foods high in fat, starches or sugars, 5) limited consumption of red and processed meat, 6) limited consumption of sugar-sweetened drinks, 7) low alcohol consumption and 8) non-smoking. The healthy lifestyle score thus ranges from 0 (worst, meaning no compliance to health recommendations) to 8 points (best, meaning full compliance to health recommendations).

SECONDARY OUTCOMES:
Participation in colorectal cancer screening | Within 6 months after sending of the faecal screening test kit to the participant at first screening round
  Return of the faecal screening test sample to the laboratory in ColorectalScreen Norway. Participants receive status 1 if a faecal screening sample is registered at the laboratory, and 0 if a faecal screening sample is not registered at the laboratory.
Completion of the Digikost questionnaire at baseline | Within 3 months after receiving the invitation to the study
  Participant invited to the trial registers him/herself at the digital study platform and fills in the first round Digikost questionnaire. Participants receive status 1 if completing, and 0 if not completing the questionnaire at baseline.
Long-term cancer incidence | From enrollment to the end of follow-up at 16 years
  Incidence of any cancer site registered in Cancer Registry after enrollment to the study. The outcome measure includes the ICD code of the diagnosis and the date of diagnosis.
Long-term cancer-specific mortality | From enrollment to the end of follow-up at 16 years
  Any cancer site as the death cause registered in Cancer Registry after enrollment to the study. The outcome measure includes the ICD code of the death cause and date of death.
Long-term total mortality | From enrollment to the end of follow-up at 16 years
  Death of any cause registered in the Death Cause Registry after enrollment to the study. The measure includes the ICD code of death cause and date of death.
Acceptability | Baseline and 1 month
  Acceptability refers to how well the Digikost questionnaire and the intervention will be received by the screening population and the extent to which the intervention is perceived as motivating in the target population. Acceptability will be assessed through qualitative interviews with participants to explore their perceptions with the intervention.
Feasibility of conducting the study, retention | 6, 12, 18 and 24 months
  Feasibility refers to how feasible it is to conduct the study. Feasibility will be assessed by participation rate in the Digikost questionnaire at repated rounds after the baseline. Participants receive status 1 if completing, and 0 if not completing the questionnaire.
Feasibility of conducting the study, attendance in the personal consultation telephone meetings | Baseline
  Feasibility refers to how feasible it is to conduct the study. Feasibility in the "High intensity lifestyle advice" group will be assessed by participation rate in the personal consultation telephone meetings at baseline. Participants receive status 1 if having completed a telephone meeting, and 0 if not having completed a telephone meeting.
Feasibility of conducting the study, attendance in the motivational webinars | 6, 12, 18 and 24 months
  Feasibility refers to how feasible it is to conduct the study. Feasibility in the "High intensity lifestyle advice" group will be assessed by participation rate in the webinars every 6 months. Participants receive status 1 if having joined a webinar, and 0 if not having not having joined a webinar.

CONTACTS AND LOCATIONS:
Overall Officials: Anette Hjartåker, PhD, Principal Investigator — University of Oslo
Locations (1):
- Norwegian Institute of Public Health, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
The ethical approval for the data ownership is limited to the study group.

REFERENCES:
- See also: Website for the project at University of Oslo — https://www.med.uio.no/imb/english/research/projects/koloprev/index.html
- See also: Website for the project at the Norwegian Institute of Public Health — https://www.fhi.no/cristin-prosjekter/aktiv/koloprev---et-randomisert-forsok-for-fokus-pa-levevaner-i-tarmscreeningprogram/